CLINICAL TRIAL: NCT06144138
Title: Impact of Breathing Exercises and Meditation on Reducing Stress and Improving Quality of Life of Glaucoma Patients: An Electronic Pilot Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 124123
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma; Stress; Quality of Life
Keywords: Glaucoma; Breathing; Meditation; Stress; Quality of life; Future consequences
MeSH Terms: conditions — Glaucoma; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercises followed by Meditation (Experimental): Breathing exercises and Meditation taught by Prasanna Wellness, a non-profit organization, helps dissolve stress and create a proper system in the mind. These breathing exercises include slow deep breaths and rapid breaths and are followed by meditation. Participants will receive three weekly online instructions (90 minutes each) by trained instructors in addition to standard care. Weekly 60 minutes follow-ups will include 10 minutes of breathing exercises followed by 33 minutes of guided meditation practice, and then focus on participants' experiences with breathing exercise followed by meditation during the week, additional observations, and a review of relevant knowledge to support their home practice.
  Interventions: Behavioral: Breathing Exercises followed by Meditation
- Treatment as Usual (No Intervention): The usual standard of care for patients with glaucoma includes starting them on first line of drugs. Participants will be initiated and maintained on appropriate dosages of such medications as part of standard of care. The usual standard of care also includes an ophthalmic examination measuring best-corrected Snellen VA and pinhole acuities and a follow-up visit once a year.

INTERVENTIONS:
Behavioral: Breathing Exercises followed by Meditation — Breathing exercises and Meditation taught by Prasanna Wellness, a non-profit organization, helps dissolve stress and create a proper system in the mind. These breathing exercises include slow deep breaths and rapid breaths and are followed by meditation. Meditation is a guided meditation that helps to eliminate stress and establish an apposite system in the mind, therefore inducing physiological and mental relaxation whilst the eyes are shut. The proposed duration and frequency of the follow-up will be 60-minutes weekly for 11 weeks.
  Arms: Breathing Exercises followed by Meditation

SUMMARY:
The goal of this electronic feasibility clinical trial study is to evaluate the effects of breathing and meditation techniques on stress levels in patients with glaucoma.

The main questions it aims to answer are:

* Does breathing and meditation decrease the level of stress in glaucoma patients?
* Does breathing and meditation improve disease specific quality of life in glaucoma patients
* Does breathing and meditation affect the importance that in glaucoma patients place on future consequences? Participants will participate in online session where they will be taught proper breathing and meditation technique to practice. They will also be completing online questionnaires following independent practice sessions over time.

Researchers will compare the breathing and meditation group to the usual care group to see if the outcomes are different.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with glaucoma. Being able to provide valid informed consent to participate in the research study.

Patients aged 40-65. Being able to read and understand English. Having no significant self-reported or physician-diagnosed mental health disorder.

Independent access to a computer to participate in virtual sessions. Must be able to sit comfortably for 30-35 minutes without any major pain or discomfort, can hear well enough to follow verbal instructions when the eyes are closed, and be in good general physical health.

Exclusion Criteria:

Inability to provide valid informed consent. Significant communication barriers or lack of English proficiency that prevents participants from completing the questionnaires.

Having a lifetime diagnosis of self-reported other serious mental disorders, including bipolar I or II disorder, primary psychotic disorder (schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder).

Self-reported substance abuse or dependence within the past 3 months. Having acutely unstable medical illnesses, including delirium or acute cerebrovascular or cardiovascular events within the last 6 months.

Having irreversible vision loss that prevents one from completing the questionnaires.

Participation in a study involving similar techniques.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life (QoL) | Baseline visit, Week 1, Week 3, Week 6, Week 12
  QoL helps physician identify hidden morbidity in clinical care as well as improves patient-physician communications. QoL will be measured using the 15-item Glaucoma Quality of Life (GQL-15) survey.
  The total score can range from 15 to 75, with higher scores indicating a poorer quality of life and a greater impact of glaucoma on one's well-being, and lower scores indicating a better quality of life and less impact of glaucoma on one's well-being.
Change in Perceived Stress | Baseline visit, Week 1, Week 3, Week 6, Week 12
  Perceived stress refers to an individual's subjective assessment of the level of stress they experience in response to various life events or circumstances.10-item Perceived Stress Scale (PSS-10).
  The total score can range from 0 to 40, with higher scores indicating higher perceived stress levels and greater psychological distress, while lower scores indicate lower perceived stress levels and less psychological distress.
Change in consideration of future consequences | Baseline visit, Week 1, Week 3, Week 6, Week 12
  Consideration of Future Consequences scale (CFC-10). The total score can range from 10 to 50, with higher scores indicating a stronger consideration of future consequences in decision-making and a greater tendency to prioritize long-term outcomes over short-term rewards, while lower scores suggest a weaker consideration of future consequences and a greater focus on immediate gratification and short-term benefits.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) collected in this study will not be available to other researchers (e.g., outside the primary research group). Since the primary research group has the necessary expertise to analyze the data and do not need any outside help.